CLINICAL TRIAL: NCT01377077
Title: Autologous Punch Grafting in Vitiligo Patients: the Effect of Punchdepth and Punchsize
Brief Title: Punchgrafting Techniques for Vitiligo
Acronym: MiniSNIP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Albert Wolkerstorfer, MD PhD, Netherlands Institute for Pigmentdisorders
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SNIP punchgrafting study
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Non-segmental Vitiligo; Segmental Vitiligo; Piebaldism
Keywords: vitiligo; piebaldism; punchgrafting; minigrafting; stable for at least 12 months
MeSH Terms: conditions — Piebaldism; Vitiligo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- epidermal 1mm grafting (Experimental): Epidermal skin biopsies of 1mm diameter
  Interventions: Procedure: punchgrafting
- dermal 1mm grafting (Experimental): dermal skinbiopsies of 1mm diameter
  Interventions: Procedure: punchgrafting
- dermal 1,5mm grafting (Experimental): dermal skinbiopsies of 1,5mm diameter
  Interventions: Procedure: punchgrafting
- epidermal 1,5mm grafting (Active Comparator): epidermal skinbiopsies of 1,5mm diameter
  Interventions: Procedure: punchgrafting

INTERVENTIONS:
Procedure: punchgrafting — autologous skin transplantation of small skinbiopsies taken from the hip and replaced in the depigmented lesions
  Arms: dermal 1mm grafting; epidermal 1,5mm grafting; epidermal 1mm grafting
Procedure: punchgrafting — autologous skingrafting of small skin biopsies taken from the hip en placed in the depigmented lesions

SUMMARY:
Rationale: Punch grafting is a safe, simple and widely used technique for in vitiligo. However, no reliable data are available on the effect of punch depth and punch size.

Objectives: Primary: to compare the efficacy and safety of different punchdepths and punchsizes in punch grafting in patients with segmental and non-segmental vitiligo. Secondary: to assess the practical aspects and patients preference of different punch grafting techniques.

Study design: Prospective observer blinded randomised controlled study. Study population: 35 patients ≥ 18 years with segmental or stable non-segmental vitiligo who will receive regular treatment by punch grafting at the Netherlands Institute for Pigment Disorders (SNIP) at the Academic Medical Centre University of Amsterdam.

Methods: Four depigmented regions on the trunk or upper extremities will be randomly allocated to either epidermal 1,5 mm punch grafting, epidermal 1mm punch grafting, dermal 1,5 mm punch grafting and dermal 1 mm punch grafting. After grafting, all regions will receive UV-therapy twice a week for 3 months. Three and six months after grafting, the repigmentation of the lesions will be assessed by measuring the outgrowth.

Main study parameter/endpoint: Outgrowth of pigment after six months.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study involves 16 additional punch grafts but no additional visits to our institute. Patients will not miss any regular treatment. The extra time due to participation in the study will be about 40 minutes. No increase of the risk of side effects is expected by placing 16 additional punch grafts. 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental and segmental vitiligo under medical treatment at the Netherlands Institute for Pigment Disorders
* Age between 18 and 60 years
* Patient is willing and able to give written informed consent
* Vitiligo stable since 12 months without systemic therapy or 6 months without topical therapy as defined by the absence of new lesions and/or enlargement of existing lesions.
* Vitiligo lesions on the extremities or trunk larger than 5x5cm

Exclusion Criteria:

* UV therapy or systemic immunosuppressive treatment during the last 12 months
* Local treatment of vitiligo during the last 6 months
* Vitiligo lesions with folliculair or non-folliculair repigmentations
* Skin type 1
* Hypertrophic scars
* Keloid
* Cardial insufficiency
* Patients with a history of hypersensitivity to (UVB) light and allergy to local anesthesia.
* Patients who are pregnant or breast-feeding
* Patients not competent to understand what the procedures involved
* Patients with a personal history of melanoma or non-melanoma skin cancer
* Patients with a first degree relative with melanoma skin cancer
* Patients with atypical nevi.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Outgrowth of pigment after six months | at 3 and 6 months after treatment
  Objective assessment of the repigmentation 3 and 6 months after punch grafting. Assessment will be done using a ruler on a dermatoscope to measure the diameter of the growth of the punchgrafts. The surface of repigmentation will be calculated.

SECONDARY OUTCOMES:
Visual assessment of side effects | at 3 and 6 months after treatment
  Visual assessment of side effects (hyperpigmentation, hypopigmentation, scar, cobble stone effect on a scale from 0-3) by a blinded investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Institute for Pigmentdisorders, Amsterdam, North Holland, Netherlands